CLINICAL TRIAL: NCT04413578
Title: Assessing the Feasibility of Continuous Glucose Monitoring in Reimagine Primary Care Clinics
Brief Title: CGM - Reimagine Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1050955
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Continuous Glucose Monitor (CGM); Dexcom G6
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Control Trial
Masking Description: Patients were either randomized to the Dexcom G6 Device or the Contour NextOne a Standard of Care glucometer. Both subjects knew what they received after they were randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dexcom G6 (Intervention Group) (Experimental): • Intervention group: CGM using a Dexcom G6 to measure glycosylated hemoglobin levels every five minutes. Patients will be asked to download the Dexcom G6 and Clarity applications (to have access to their real-time data) and be given a link to complete an exit survey in REDCap near the end of their study participation. Data will be sent via Bluetooth and then exported by the Intermountain research team into a Tableau (or similar) dashboard for data analysis/comparison
  Interventions: Device: Dexcom G6
- Contour NextOne (Standard of Care) Glucometer (Placebo Comparator): • Control group: A standard finger-prick protocol that will require patients to continue with their daily fingerprick regimen established by their physician. This group will be given a Contour Next One meter to ensure that each patient is receiving the same level of accuracy by the same device. A review by Ekhlaspour et al of 17 glucose meters demonstrated wide variability, with only two devices achieving the 2013 ISO standard (with the most accurate being the Contour Next). Patients in the control group will be asked to download the Contour Next application which will send data via Bluetooth similar to above. Data will be aggregated, and protected health information removed prior to analysis (by Intermountain Healthcare and Savvysherpa). At the end of the study, patients will be asked to complete a short survey in REDCap about their willingness to participate in future studies.
  Interventions: Device: Contour NextOne

INTERVENTIONS:
Device: Dexcom G6 — Continuous Glucose Monitor that, after applied, sends continuous glucose readings to to the patient's smartphone every 5 minutes. This allows the patients to receive more readings over a 24 hour period versus standard of care glucometer finger sticks.
  Arms: Dexcom G6 (Intervention Group)
Device: Contour NextOne — A Standard of Care Glucometer with Bluetooth capability. The patient inserts a test strip into the device, takes a finger stick and collects a small blood sample on the tip of the strip to initiate the device to detect a glucose reading.
  Arms: Contour NextOne (Standard of Care) Glucometer

SUMMARY:
To assess the impact of continuous glucose monitoring versus standard of care (e.g. a finger-prick protocol using a glucometer) on clinical outcomes, healthcare utilization, and cost in patients with type I or II diabetes treated within the Reimagine Primary Care clinics.

DETAILED DESCRIPTION:
This is a parallel randomized controlled trial. Eligible patients who consent will be randomized to one of two groups: (1) the intervention group who will be given a Dexcom G6 for CGM, or (2) the control group who will follow their current standard finger-prick protocol via a provided Contour Next ONE glucometer. The CGM group must download the Dexcom G6 and Clarity mobile apps for data capture, whereas the standard of care group will use the Contour Next mobile app for their respective readings.

The Dexcom G6 captures real-time, dynamic glucose data every five minutes. Devices used in this study are FDA approved and commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus with a HbA1c ≥6.5%
* Patients that are currently managing their glucose levels for diabetes with a glucose meter (or will be prescribed one by their healthcare provider)
* Patients that are treated within the four Reimagine Primary Care clinics (Cottonwood Family Medicine, Cottonwood Senior, Avenues Internal Medicine, and Holladay Internal Medicine). • Patients 18-80 years of age

Exclusion Criteria:

* Patients that are not managing their glucose levels for diabetes (and not advised to use a glucose monitor by their physician)
* Patients that are not treated within the four Reimagine Primary Care clinics
* Patients less than 18 years of age, and 81 years of age and older
* Patients with a diagnosis of dementia
* If the patient is currently using a Continuous Glucose Monitor
* Patients with previous hospitalization for hypoglycemia within the last 18 months
* No access to a mobile phone to download the Dexcom or Contour Next applications
* Patients who are pregnant or planning to become pregnant over the course of their six-month participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c Variation | 6 months
  Coefficient of variation in HbA1c levels before, during and end of study completion.
HbA1c Range | 6 months
  Variation of range in HbA1c levels before, during and end of study completion.

SECONDARY OUTCOMES:
Current Diabetes Standards | 6 months
  Current HEDIS performance on diabetes and behavioral health measures.
Behavioral Changes | 6 months
  Subjects will complete a self reported survey related to behavioral changes at end of study to assess self empowered behavioral changes after using the devices (e.g. feeling more empowered to self-manage care, engaged with changing healthcare behaviors, and patient perceptions of the technology).
Hypoglycemic Events | 6 months
  Frequency of hypoglycemic events during the study.
Healthcare Utilization | 6 months
  Healthcare utilization per count of inpatient/outpatient visits.
Glycemic Variability | 6 months
  Glycemic variability per mean amplitude of glycemic excursion (MAGE)
Emergency Room Visits | 6 months
  Emergency department visits per 1000 rate, overall and for patients with diabetes, and hospitalization per 1000 rate related to.
Healthcare Cost | 6 months
  Cost per patient of healthcare for Emergency Room visits, blood draws, inpatient/outpatient services, medications etc.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Holladay Internal Medicine, Holladay, Utah
  - Intermountain Cottonwood Family Practice, Murray, Utah
  - Intermountain Senior Clinic, Murray, Utah
  - Avenues Internal Medicine, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee PA, Greenfield G, Pappas Y. The impact of telehealth remote patient monitoring on glycemic control in type 2 diabetes: a systematic review and meta-analysis of systematic reviews of randomised controlled trials. BMC Health Serv Res. 2018 Jun 26;18(1):495. doi: 10.1186/s12913-018-3274-8. PMID 29940936
- [Result] Medical Advisory Secretariat. Home telemonitoring for type 2 diabetes: an evidence-based analysis. Ont Health Technol Assess Ser. 2009;9(24):1-38. Epub 2009 Oct 1. PMID 23074529
- [Result] Ekhlaspour L, Mondesir D, Lautsch N, Balliro C, Hillard M, Magyar K, Radocchia LG, Esmaeili A, Sinha M, Russell SJ. Comparative Accuracy of 17 Point-of-Care Glucose Meters. J Diabetes Sci Technol. 2017 May;11(3):558-566. doi: 10.1177/1932296816672237. Epub 2016 Oct 3. PMID 27697848
- [Result] Verkuilen J. Explanatory Item Response Models: A Generalized Linear and Nonlinear Approach by P. de Boeck and M. Wilson and Generalized Latent Variable Modeling: Multilevel, Longitudinal and Structural Equation Models by A. Skrondal and S. Rabe-Hesketh. Psychometrika. 2006 Jun;71(2):415-418. doi: 10.1007/s11336-005-1333-7. No abstract available. PMID 28197954
- [Result] Fong Y, Rue H, Wakefield J. Bayesian inference for generalized linear mixed models. Biostatistics. 2010 Jul;11(3):397-412. doi: 10.1093/biostatistics/kxp053. Epub 2009 Dec 4. PMID 19966070
- [Result] Musio M, Sauleau EA, Augustin NH. Resources allocation in healthcare for cancer: a case study using generalised additive mixed models. Geospat Health. 2012 Nov;7(1):83-9. doi: 10.4081/gh.2012.107. PMID 23242683
- See also: What is Diabetes — http://www.niddk.nih.gov/health-information/diabetes/overview/what-is-diabetes
- See also: Diabetes and glucose information — http://professional.diabetes.org/diapro/glucose_calc

DOCUMENTS (2):
  • Informed Consent Form (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT04413578/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT04413578/Prot_SAP_001.pdf